CLINICAL TRIAL: NCT02414165
Title: A Phase 2/3 Randomized, Open-Label Study of Toca 511, a Retroviral Replicating Vector, Combined With Toca FC Versus Standard of Care in Subjects Undergoing Planned Resection for Recurrent Glioblastoma or Anaplastic Astrocytoma
Brief Title: The Toca 5 Trial: Toca 511 & Toca FC Versus Standard of Care in Patients With Recurrent High Grade Glioma
Acronym: Toca5
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-15-01; FD-R-5732 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2015-04-03; First posted 2015-04-10 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: Recurrence
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Recurrence | interventions — vocimagene amiretrorepvec; Flucytosine; Lomustine; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toca 511/Toca FC (Experimental): Resection followed by administration of 4 mL Toca 511 (vocimagene amiretrorepvec). Toca 511 is administered by injection into the wall of the subject's tumor resection cavity on Day 1 (approximately 40 injections of 0.1 mL)
  Toca FC is an extended-release formulation of flucytosine. Toca FC will be administered at 220 mg/kg/day orally for 7-day courses beginning at least 6 weeks after resection and repeated approximately every 6 weeks.
  Interventions: Biological: Toca 511; Drug: Toca FC
- Lomustine, Temozolomide, or Bevacizumab (Active Comparator): Investigator selects one of the following:
  Bevacizumab: Beginning 6 weeks after tumor resection, bevacizumab will be administered by IV infusion at 10 mg/kg and repeated every 2 weeks. Refer to the prescribing information and to institutional guidelines for details on the administration procedure.
  Lomustine: Beginning 6 weeks after tumor resection, lomustine will be administered as a single oral dose of 110 mg/m2 and repeated every 6 weeks. Refer to the prescribing information and to institutional guidelines for details regarding the administration procedure.
  Temozolomide: Beginning 6 weeks after tumor resection, temozolomide will be administered per 1 of 2 options:
  * at a dose of 50 mg/m2 PO once daily continuously, or
  * at an initial dose of 150 mg/m2 IV or PO once daily for 5 consecutive days per 28-day treatment cycle that may be raised to 200 mg/ m2 once daily for 5 consecutive days in the following 28-day treatment cycles
  Interventions: Drug: Lomustine; Drug: Temozolomide; Biological: Bevacizumab

INTERVENTIONS:
Biological: Toca 511 — Toca 511 consists of a purified retroviral replicating vector encoding a modified yeast cytosine deaminase (CD) gene. The CD gene converts the antifungal 5-flurocytosine (5FC) to the anticancer drug 5-FU in cells that have been infected by the Toca 511 vector.
  Other Names: vocimagene amiretrorepvec; RRV; retroviral replicating vector
  Arms: Toca 511/Toca FC
Drug: Toca FC — Toca FC is an extended-release formulation of flucytosine and is supplied as 500 mg tablets
  Other Names: flucytosine; 5-FC; 5-fluorocytosine
  Arms: Toca 511/Toca FC
Drug: Lomustine
  Other Names: CCNU; CeeNU
  Arms: Lomustine, Temozolomide, or Bevacizumab
Drug: Temozolomide
  Other Names: Temodar
  Arms: Lomustine, Temozolomide, or Bevacizumab
Biological: Bevacizumab
  Other Names: Avastin
  Arms: Lomustine, Temozolomide, or Bevacizumab

SUMMARY:
This is a multicenter, randomized, open-label phase 2/3 study of Toca 511 and Toca FC versus standard of care that comprises Investigator's choice of single agent chemotherapy (lomustine or temozolomide) or bevacizumab administered to subjects undergoing resection for first or second recurrence (including this recurrence) of GBM or AA. Subjects meeting all of the inclusion and none of the exclusion criteria will be randomized prior to surgery in a 1:1 ratio to receive either Toca 511 and Toca FC (Experimental arm, Arm T) or control treatment with one option of standard of care (Arm SOC). Stratification will be done by IDH1 mutation status. A second stratification factor is based on the patient's Karnofsky Performance Score (KPS) (70-80 vs 90-100). Further, to account for potential differences in treatment choices for the control arm in regions, the trial will be stratified by geographical region during the randomization process.

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Subject is between 18 years old and 75 years old, inclusive
3. Subjects must have histologically proven GBM or AA and:

   1. Must have received first-line multimodal therapy with surgery followed by temozolomide (unless MGMT promoter unmethylated) and radiation (subjects with GBM must have received temozolomide and radiation concurrently)
   2. Must be in first or second recurrence (including this recurrence)
   3. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI. If first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field
4. Subjects must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per RANO criteria
5. Subjects must be at least 4 weeks post last dose of temozolomide
6. Prior gamma knife, stereotactic radiosurgery, or other focal high-dose radiotherapy is allowed but the subject must have either histopathologic confirmation of recurrent tumor, or new enhancement on MRI outside of the radiotherapy treatment field
7. Based on the pre-operative evaluation by neurosurgeon, the subject is a candidate for ≥ 80% resection of enhancing region
8. IDH mutation status of the primary tumor must be available or tumor samples must be available for pre randomization testing
9. Laboratory values adequate for patient to undergo surgery, including:

   * Platelet count ≥ 60,000/mm3
   * Hgb ≥ 10 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Absolute lymphocyte count (ALC) ≥ 500/mm3
   * Adequate liver function, including:

     * Total bilirubin ≤ 1.5 x ULN (unless has Gilbert's syndrome)
     * ALT ≤ 2.5 x ULN f. Estimated glomerular filtration rate of at least 50 mL/min by the Cockcroft Gault formula
10. Women of childbearing potential (≥12 months of non-therapy-induced amenorrhea or surgically sterile) must have had a negative serum pregnancy test within the past 21 days and must use a birth control method in addition to barrier methods (condoms).
11. Subject or subject's partner is willing to use condoms for 12 months after receiving Toca 511 or until there is no evidence of the virus in his/her blood, whichever is longer.
12. The subject has a KPS ≥ 70
13. The subject is willing and able to abide by the protocol

Exclusion Criteria:

1. History of more than 2 prior recurrences (including this recurrence) of GBM or AA
2. History of other malignancy, unless the patient has been disease free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment
3. Histologically confirmed oligodendroglioma or mixed glioma
4. Known 1p/19q co deletion
5. A contrast enhancing brain tumor that is any of the following:

   * Multi focal (defined as 2 separate areas of contrast enhancement measuring at least 1 cm in 2 planes that are not contiguous on either fluid attenuated inversion recovery (FLAIR) or T2 sequences);
   * Associated with either diffuse subependymal or leptomeningeal dissemination; or
   * > 5 cm in any dimension
6. The subject has or had any active infection requiring systemic antibiotic, antifungal or antiviral therapy within the past 4 weeks
7. The subject has any bleeding diathesis, or must take anticoagulants, or antiplatelet agents, including nonsteroidal anti inflammatory drugs (NSAIDs), at the time of the scheduled resection that cannot be stopped for surgery
8. The subject is human immunodeficiency virus (HIV) positive
9. The subject has a history of allergy or intolerance to flucytosine
10. The subject has a gastrointestinal disease that would prevent him or her from being able to swallow or absorb flucytosine
11. The subject received cytotoxic chemotherapy within the past 4 weeks (6 weeks for nitrosoureas) of the planned surgery date
12. The subject received any investigational treatment within the past 30 days or prior immunotherapy or antibody therapy within the past 45 days.
13. The subject is pregnant or breast feeding
14. The subject intends to undergo treatment with the Gliadel® wafer at the time of this surgery or has received the Gliadel® wafer < 30 days from W1D1 (surgery)
15. The subject has received bevacizumab for their disease unless in the context of primary therapy for newly diagnosed glioma
16. For subjects planned to potentially receive bevacizumab, they have no evidence of uncontrolled hypertension (defined as a blood pressure of ≥ 150 mm Hg systolic and/or ≥ 100 mm Hg diastolic on medication) or active GI perforation
17. The subject has received systemic dexamethasone continuously at a dose > 8 mg/day for 8 weeks prior to the date of the screening assessment
18. Severe pulmonary, cardiac or other systemic disease, specifically:

    * New York Heart Association > Grade 2 congestive heart failure within 6 months prior to study entry, unless asymptomatic and well controlled with medication
    * Uncontrolled or significant cardiovascular disease, clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades des pointes), clinically significant pulmonary disease (such as ≥ Grade 2 dyspnea, according to CTCAE 4.03)
    * Subjects who have any other disease, either metabolic or psychological, which as per Investigator assessment may affect the subject's compliance or place the subject at higher risk of potential treatment complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
To compare the overall survival (OS) of subjects treated with Toca 511 combined with Toca FC to subjects treated according to standard of care after tumor resection for recurrence of glioblastoma or anaplastic astrocytoma | 30 December 2019
  Time from randomization date to death due to any cause

SECONDARY OUTCOMES:
Durable Response Rate (CR or PR ≥ 24 weeks) | 30 December 2019
  The proportion of patients whose best response is either CR or PR lasting at least 24 weeks, according to modified RANO criteria
Durable Clinical Benefit Rate (CR or PR ≥ 24 weeks or SD ≥ 18 months) | 30 December 2019
  The proportion of subjects whose best overall response is either CR or PR lasting at least 24 weeks, or stable disease (SD) lasting at least 18 months, according to modified RANO criteria
Duration of Durable Response | 30 December 2019
  Time from documentation of durable response to disease progression or death due to disease progression
Overall Survival at 12 months | 30 December 2019
  Time from randomization date to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cloughesy, MD, Principal Investigator — University of California, Los Angeles
Locations (67):
- United States (50):
  - Barrow Neurological Institute at Dignity Health St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of California San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - St. Joseph Hospital, Orange, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Yale University/Yale Cancer Center, New Haven, Connecticut
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - NorthShore University Health System, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Abbott Northwestern Hospital / Allina Health, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - HCA Midwest / Sarah Cannon, Kansas City, Missouri
  - Washington University St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - JFK Medical Center Neuroscience Institute, Edison, New Jersey
  - John Theurer Cancer Center at Hackensack University, Hackensack, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - North Shore University Hospital, Lake Success, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Cincinnati's Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital Outpatient Center, Houston, Texas
  - University of Texas Health Science Center at Houston (UTHealth), Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Dwight and Martha Schar Cancer Institute, Fairfax, Virginia
  - Sentara Neurosurgery Specialists, Norfolk, Virginia
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (10):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia / Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Hospital / Sunnybrook Research Institute, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Sherbrooke Hospital University Centre (CHUS), Sherbrooke, Quebec
- Israel (3):
  - Rambam Health Care, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

REFERENCES:
- [Derived] Cloughesy TF, Petrecca K, Walbert T, Butowski N, Salacz M, Perry J, Damek D, Bota D, Bettegowda C, Zhu JJ, Iwamoto F, Placantonakis D, Kim L, Elder B, Kaptain G, Cachia D, Moshel Y, Brem S, Piccioni D, Landolfi J, Chen CC, Gruber H, Rao AR, Hogan D, Accomando W, Ostertag D, Montellano TT, Kheoh T, Kabbinavar F, Vogelbaum MA. Effect of Vocimagene Amiretrorepvec in Combination With Flucytosine vs Standard of Care on Survival Following Tumor Resection in Patients With Recurrent High-Grade Glioma: A Randomized Clinical Trial. JAMA Oncol. 2020 Dec 1;6(12):1939-1946. doi: 10.1001/jamaoncol.2020.3161. PMID 33119048
- [Derived] Cloughesy TF, Landolfi J, Hogan DJ, Bloomfield S, Carter B, Chen CC, Elder JB, Kalkanis SN, Kesari S, Lai A, Lee IY, Liau LM, Mikkelsen T, Nghiemphu PL, Piccioni D, Walbert T, Chu A, Das A, Diago OR, Gammon D, Gruber HE, Hanna M, Jolly DJ, Kasahara N, McCarthy D, Mitchell L, Ostertag D, Robbins JM, Rodriguez-Aguirre M, Vogelbaum MA. Phase 1 trial of vocimagene amiretrorepvec and 5-fluorocytosine for recurrent high-grade glioma. Sci Transl Med. 2016 Jun 1;8(341):341ra75. doi: 10.1126/scitranslmed.aad9784. PMID 27252174